CLINICAL TRIAL: NCT00672321
Title: Melanoma Lifestyle Study
Brief Title: Answering Questions About Vitamin D Supplementation and Sun Exposure in Patients Who Have Undergone Surgery for Stage IB, Stage II, or Stage IIIA Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leeds Cancer Centre at St. James's University Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: LCC-MREC-07-H1010-66; CDR0000587987 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-05-03; First posted 2008-05-06 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IB melanoma; stage II melanoma; stage IIIA melanoma
MeSH Terms: conditions — Melanoma | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Gathering information about vitamin D supplementation and sun exposure in patients with melanoma may help doctors learn more about the disease and find what may affect cancer relapse.

PURPOSE: This clinical trial is studying vitamin D supplementation and sun exposure in patients who have undergone surgery for stage IB, stage II, or stage IIIA melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To examine the findings of the pilot study, that vitamin D supplementation in combination with vitamin D receptor (VDR) polymorphisms protects from late relapse (after 3 years) in patients who have had melanoma.
* To investigate the effects of vitamin D supplement dosage in reducing the risk of late relapse.
* To examine if vitamin D supplementation in combination with particular VDR polymorphisms protects from early relapse (before 3 years).
* To examine if serum levels of vitamin D correlate with risk of relapse in groups of patients with different VDR polymorphisms.
* To examine the effect of vitamin supplementation and VDR status on time to relapse and survival in these patients.
* To examine other factors that may affect risk of relapse by assembling a tissue (genomic DNA and serum) resource.
* To investigate the effect of exposure to incidental drugs, such as statins, on risk of relapse in these patients.

OUTLINE: Patients are stratified according to disease relapse in the past 5 years (yes vs no).

Patients are asked to complete a food frequency questionnaire focusing on vitamin D and the following area: supplementation of diet with vitamins/fish oil and duration of use; sun exposure and sunscreen-use per decade prior to and after diagnosis. Patients are also asked to provide a blood sample for serum and DNA analysis. Consenting patients are also tagged with the Office of National Statistics to allow passive follow up.

Stored tissue from the patient's primary melanoma may be used to corroborate research findings using immunohistochemistry or studies of gene expression, polymorphism, or mutation.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with melanoma
* Must meet either of the following conditions:

  * Resected stage IB, II, or IIIA disease that has relapsed as either stage III or IV disease (cases)

    * First loco regional and/or visceral relapse (with/without sentinel node biopsy)

      * No more than 3 months since first relapse
  * Resected stage IB, II, or IIIA disease that has not relapsed for ≥ 5 years (controls)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2774 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Odds ratio (OR) for vitamin D supplementation in relapse
OR for vitamin D supplementation in patients with specific VDR genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Julia Newton Bishop, MD, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom